CLINICAL TRIAL: NCT07194005
Title: Efficacy and Safety of RC48 (Disitamab Vedotin) Combined With Sintilimab and SOX for HER2 IHC 1+/2+ Unresectable Locally Advanced or Advanced Gastric Cancer Conversion Therapy
Brief Title: Conversion Therapy With RC48, Sintilimab, and SOX for HER2 1+/2+ Unresectable Gastric Cancer
Acronym: Remission
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fenglin Liu, Director of Gastric Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC092
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; disitamab vedotin; conversion therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Disitamab vedotin in combination with sintilimab and SOX as conversion therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion therapy (Experimental): Drug: Disitamab Vedotin in combination with sintilimab and SOX
  Interventions: Drug: Disitamab vedotin(RC48); Drug: Sintilimab; Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Disitamab vedotin(RC48) — 2.5 mg/kg, administered intravenously every 3 weeks (Q3W) on Day 1 of each cycle.
  Other Names: RC48
Drug: Sintilimab — 200 mg, administered intravenously, d1, every 3 weeks.
Drug: S-1 — Oral, 40-60 mg, twice daily (bid), d1-14, every 3 weeks.
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule
Drug: Oxaliplatin — 130 mg/m², administered intravenously on Day 1 (d1), every 3 weeks.

SUMMARY:
This study aims to evaluate the efficacy of disitamab vedotin in combination with sintilimab and SOX as conversion therapy in patients with initially unresectable locally advanced or metastatic gastric cancer exhibiting HER2 IHC 1+/2+ expression. The trial plans to enroll patients with a single initial unresectable factor and HER2 IHC 1+/2+ status. Participants will receive disitamab vedotin combined with sintilimab and SOX for 4 to 6 treatment cycles. Those who achieve successful conversion will undergo surgical resection, while patients with unsuccessful conversion will either continue the original regimen or switch to an alternative treatment at the investigator's discretion.

DETAILED DESCRIPTION:
This is an open-label, single-arm, exploratory study designed to enroll patients with a single initial unresectable factor and HER2 IHC 1+/2+ locally advanced or metastatic gastric cancer. The primary objective is to assess the efficacy of the combination regimen based on the R0 resection rate. Tumor response will be evaluated every 6 to 12 weeks via imaging to determine whether surgical criteria are met. Patients who meet the criteria for operability will proceed to surgery, and postoperative adjuvant therapy will be tailored by the investigator based on individual patient conditions. For those who do not achieve successful conversion, the investigator will decide whether to continue the original treatment or transition to an alternative therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily enrolled and provided written informed consent;
2. Aged 18-70 years (inclusive), male or female;
3. Histologically and/or cytologically confirmed unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma;
4. No prior systemic anticancer therapy;
5. HER2 immunohistochemistry (IHC) result of 2+ or 1+, based on either previous test results (confirmed by the investigator) or central laboratory assessment;
6. Presence of a single initial unresectable factor;
7. At least one measurable lesion per RECIST 1.1;
8. Life expectancy ≥ 6 months;
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
10. Adequate organ function, defined as follows:

Hematological (within 14 days prior to screening, without transfusion or granulocyte colony-stimulating factor [G-CSF] support):

1. Hemoglobin ≥ 90 g/L;
2. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
3. White blood cell count ≥ 3.0 × 10⁹/L;
4. Platelet count ≥ 80 × 10⁹/L;

   Biochemical (within 14 days prior to screening, without albumin infusion):
5. Albumin ≥ 28 g/L;
6. Total bilirubin ≤ 2 × upper limit of normal (ULN);
7. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN in the absence of liver metastases; or ≤ 5 × ULN if liver metastases are present;
8. Serum creatinine ≤ 1.5 × ULN; or creatinine clearance (CrCl) ≥ 50 mL/min as calculated by the Cockcroft-Gault formula;

   Coagulation:
9. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN;
10. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

Exclusion Criteria:

1. History of malignancies other than gastric cancer, with the following exceptions:

   1. Malignancies treated with curative intent and with no evidence of disease for 5 years;
   2. Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, or other in situ carcinomas.
2. Conditions affecting the absorption, distribution, metabolism, or excretion of the investigational drug(s) (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, malabsorption, etc.).
3. Previous allogeneic stem cell or solid organ transplantation.
4. Prior systemic antitumor therapy (including Chinese herbal medicine with antitumor indications) completed less than 4 weeks before the first dose of study treatment, or with prior treatment-related adverse events not recovered to ≤ CTCAE grade 1 (except for alopecia or pigmentation).
5. History or presence of congenital or acquired immunodeficiency disorders.
6. Active or previously documented autoimmune or inflammatory disorders (including but not limited to autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, hypophysitis, hyperthyroidism, hypothyroidism, asthma requiring bronchodilators, etc.). Patients with vitiligo, childhood asthma that has fully resolved without intervention in adulthood, or other conditions deemed eligible by the investigator may be included.
7. Use of systemic immunosuppressive therapy within 2 weeks prior to enrollment, or anticipated need for such therapy during the study, with the following exceptions:

   1. Intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular);
   2. Systemic corticosteroids at a dose ≤ 10 mg/day prednisone or equivalent;
   3. Prophylactic corticosteroids for hypersensitivity reactions.
8. Known or suspected history of hypersensitivity to disitamab vedotin, anti-PD-1 agents, chimeric or humanized antibodies or fusion proteins, or any excipient of the investigational drug(s).
9. History of thrombotic or thromboembolic events within the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.
10. Patients assessed by the physician to be at significant risk of bleeding, including but not limited to:

    * Major bleeding (>30 mL within 3 months) or hemoptysis (>5 mL within 4 weeks); endoscopic evaluation may be performed to confirm eligibility;
    * Active bleeding or coagulation disorders;
    * Bleeding tendency or current use of thrombolytic, anticoagulant, or antiplatelet therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | Within 1 month of surgery
  Defined as no residue under the microscope after resection

SECONDARY OUTCOMES:
Pathologic complete response | Within 1 month of surgery.
  The number of people who have achieved complete pathological remission accounted for the proportion of people who met the plan.
Overall survival | 2 years from the start of system therapy.
  The time from the start of system therapy to the death of any cause.
1/2-year survival rate | 1/2 years from the start of system therapy.
  Percentage of subjects who are alive without death event at 1/2 years.
Adverse events(all grades） | From the start of system therapy to 6 months after surgery.
  Assessed per Common Terminology Criteria for Adverse Events(CTCAE) version 5.0
Serious adverse events(≥grade 3） | From the start of system therapy to 6 months after surgery.
  Assessed per Common Terminology Criteria for Adverse Events(CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is protected.